CLINICAL TRIAL: NCT04390139
Title: A Prospective, Double-blind, Randomized, Parallel, Placebo-controlled Pilot Clinical Trial for the Evaluation of the Efficacy and Safety of Two Doses of WJ-MSC in Patients With Acute Respiratory Distress Syndrome Secondary to Infection by COVID-19
Brief Title: Efficacy and Safety Evaluation of Mesenchymal Stem Cells for the Treatment of Patients With Respiratory Distress Due to COVID-19
Acronym: COVIDMES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BST-COVID-01
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; SARS-CoV 2; Adult Respiratory Distress Syndrome
Keywords: ARDS
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Wharton-Jelly mesenchymal stromal cells on D1 and D3
  Interventions: Drug: XCEL-UMC-BETA
- Treatment B (Placebo Comparator): Placebo on D1 and D3
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: XCEL-UMC-BETA — Administration on top of the standard administered treatment
  Other Names: WJ-MSC
  Arms: Treatment A
Other: Placebo — Administration on top of the standard administered treatment
  Arms: Treatment B

SUMMARY:
Randomized, double-blind, parallel, two-arms clinical trial to assess the efficacy and safety of 2 infusions of Wharton-Jelly mesenchymal stromal cells (day 1 and day 3, endovenously at 1E6cells/Kg per dose) in patients with moderate acute respiratory distress syndrome (ARDS) secondary to SARS-CoV-2 infection. Follow-up will be established on days 3, 5, 7, 14, 21, and 28. Long term follow-up will be performed at 3, 6 and 12 months.

DETAILED DESCRIPTION:
This is a prospective, double-blind, randomized, parallel, placebo-controlled pilot clinical trial to assess the efficacy and safety of two infusions of Wharton Jelly mesenchymal stromal cells (WJ-MSC) in patients with moderate acute respiratory distress syndrome (ARDS) secondary to SARS-CoV-2 infection. The study will enroll 30 patients who after signing the informed consent will be checked for inclusion and exclusion criteria. Patients will then be randomized (1:1) to one of the 2 treatment arms: Treatment A WJ-MSC/WJ-MSC; Treatment B Placebo/ Placebo. The 2 infusions will be administered endovenously on day 1 (D1) and on D3. Thereafter, patients will be followed-up on days 3, 5, 7, 14, 21, and 28 Once the study is completed, controls will be established at 3 months, 6 months and 12 months as long-term follow-up.

The study treatments (A or B) will be added on top of the Standard of Care treatment prescribed by the attending physician. Each dose of MSC-WJ will consist of the intravenous administration of 1E6cells/Kg.

Recruitment will be competitive for the centers participating in the study. A Data Safety and Monitoring Board (DSMB) will be established to review safety and efficacy along the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Positive PCR fpr SARS-CoV-2
2. Intensive Care Unit admission for less than 3 days
3. Moderate acute respiratory distress (Berlin criteria definition with 100 mmHg < PaO2/FiO2 ≤ 200 mmHg)
4. Male or female, aged 18 to 70 years old
5. Signed informed consent by the patient or by a legal representative (in this case, can be obtained by phone, although it must be confirmed in writing later, accepted by email)

Exclusion Criteria:

1. Expected survival less than 3 days
2. Treatment with immunosuppressive drugs (tocilizumab, sarilumab) with corticosteroids being allowed
3. Neoplastic disease either active or without complete remission
4. Immunosuppressed patients (except treatment with corticosteroids for respiratory distress)
5. Pregnant or lactating women
6. Participation in another clinical trial with an experimental drug in the last 30 days
7. Other pathologies that, in medical judgment, contraindicate participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
All-cause mortality at day 28 | Day 28
  Number of patients who died, by treatment group

SECONDARY OUTCOMES:
Safety of WJ-MSC | Day 28
  Number of patients with treatment-emergent adverse events, by treatment group
Need for treatment with rescue medication | Day 28
  Number of patients who, after the start of treatment, required rescue medication, by treatment group
Need and duration of mechanical ventilation | Day 28
  Number of days that the patient requires invasive mechanical ventilation from the start of treatment to day +28, by treatment group
Ventilator free days | Day 28
  Days after treatment in which the patient remains alive and free of invasive mechanical ventilation, per treatment group.
Evolution of PaO2 / FiO2 ratio | Day 28
  Variation of the oxygenation index (PaO2 / FiO2) with respect to the baseline value, by treatment group.
Evolution of the SOFA index | Day 28
  Variation of the score of the Sequential Organ Failure Assessment (SOFA) Index with respect to the baseline value, by treatment group.
Evolution of the APACHE II score | Day 28
  Variation of Acute Physiology and Chronic Health disease Classification System II (APACHE II) score, by treatment group.
Duration of hospitalization | Day 28
  Days of stay in the ICU from the day of admission until discharge to day 28, or date of death if earlier, by treatment group.
Evolution of markers of immune response (leucocyte count, neutrophils) | Day 28
  Variation in the count and percentage of leukocytes and neutrophils, by treatment group.
Feasibility of WJ-MSC administration | Day 28
  Feasibility will be evaluated by the time elapsed from the request of the treatment by the hospital center until the delivery date
Feasibility of WJ-MSC administration | Day 28
  Feasibility will be evaluated by the number of patients treated within 2 days of the request for treatment.
Evolution of disease biomarker: polymerase chain reaction (RT-PCR) | Day 28
  Variation in the values of the biomarker, by treatment group.
Evolution of disease biomarker: lactate dehydrogenase (LDH) | Day 28
  Variation in the values of the biomarker, by treatment group.
Evolution of disease biomarker: D-dimer | Day 28
  Variation in the values of the biomarker, by treatment group.
Evolution of disease biomarker: Ferritin | Day 28
  Variation in the values of the biomarker, by treatment group.

OTHER OUTCOMES:
Analysis of subpopulations of lymphocytes and immunoglobulins | Day 28
  Blood sample analysis
Evaluation of the in vitro response of the receptor lymphocytes | Day 28
  In vitro response will be assessed using commercial viral antigens (Miltenyi Biotech)
Study of reactivity against SARS-CoV-2 peptides | Day 28
  Reactivity will be assessed using ELISPOT
Immunophenotypic study of memory cells in response to SARS-CoV-2 peptides | Day 28
  Blood sample analysis
Genetic variability of patient's genotype in response to treatment | Day 28
  Blood sample analysis for the patient's genomic sequencing
Genetic variability of the SARS-CoV-2 genotype in response to treatment | Day 28
  Genomic sequencing of the SARS-CoV-2 in a nasopharyngeal sample

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Torres, MD, PhD, Study Chair — Hospital Clinic of Barcelona
Locations (5):
- Spain (5):
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Mútua de Terrassa, Terrassa, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Blood and Tissue Bank of Catalonia — http://www.bancsang.net
- See also: Hospital Clínic de Barcelona — http://www.clinicbarcelona.org
- See also: Hospital Vall d'Hebron — http://www.vallhebron.com
- See also: Hospital del Mar — http://www.parcdesalutmar.cat
- See also: Mútua de Terrassa — http://www.mutuaterrassa.com
- See also: Hospital de Bellvitge — http://bellvitgehospital.cat